CLINICAL TRIAL: NCT03977831
Title: A Controlled Blinded Randomized Feasibility Study of Open Radical Cystectomy (ORC) Versus Robot-Assisted Radical Cystectomy With Intracorporal Urinary Diversion (iRARC) Under an Enhanced Recovery After Surgery (ERAS) Setup
Brief Title: Study Comparing Open Radical Cystectomy With Robot-assisted Cystectomy in Patients With Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulla Nordström Joensen, Associate Professor, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-18056682-D
Record Dates: First submitted 2019-05-29; First posted 2019-06-06 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Bladder Cancer; Radical cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cystectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Radical Cystectomy (ORC) (Active Comparator): Open radical cystectomy includes in both genders removal of the bladder and distal ureters as well as pelvic lymphadenectomy. In men the procedure includes removal of the prostate and seminal vesicles and in women removal of the uterus, ovaries, urethra and part of the vagina. Lastly, for both genders an iliac conduit urinary diversion is performed.
  Interventions: Procedure: Radical Cystectomy
- Robot-assisted Radical Cystectomy (iRARC) (Active Comparator): Robot-assisted radical cystectomy includes in both genders removal of the bladder and distal ureters as well as pelvic lymphadenectomy. In men the procedure includes removal of the prostate and seminal vesicles and in women removal of the uterus, ovaries, urethra and part of the vagina. Lastly, for both genders an intracorporeal iliac conduit urinary diversion is performed.
  Interventions: Procedure: Radical Cystectomy

INTERVENTIONS:
Procedure: Radical Cystectomy — Participants are randomly and blinded assigned

SUMMARY:
The purpose of the study to compare two established methods of radical cystectomy (RC) in patients with bladder cancer. The participants will be treated under conditions in alignment with up-to-date guidelines and care. We wish to investigate whether it is feasible to compare the two methods under conditions of the highest methodological quality.

DETAILED DESCRIPTION:
Radical cystectomy (RC) is a comprehensive surgery including pelvic lymph node dissection and urinary diversion. The surgery is originally performed as an open procedure (ORC) but with advances in technology the procedure is now also offered as a robot-assisted laparoscopic procedure (RARC). It remains questionable if RARC is superior to ORC in terms of surgical outcomes.

Several studies have described outcomes following RARC of which most are comparative studies with only five studies being randomized controlled trials (RCTs). Overall, significant differences in operating room time, estimated blood loss, time to flatus and bowel movement as well as use of morphine sulfate equivalents in favor of RARC has been demonstrated with the exception of operating room time. However, no studies have demonstrated a significant reduction in risk of 30- or 90-day complication rates between ORC and RARC. The RCTs have not been blinded, and therefore may be subject to bias in terms of expectations from patients and care providers. Also, in the already conducted RCTs of ORC versus RARC the urinary diversion has been done extracorporally. Today, it is possible to conduct the whole procedure of RARC intracorporally (iRARC), potentially reducing the surgical stress further. Lastly, the previously conducted RCTs have not consequently been managed under an Enhanced Recovery After Surgery (ERAS) setup. Currently, a multicenter study comparing ORC with RARC is recruiting in the United Kingdom in which the patients are treated with iRARC and under an ERAS setup. The present study will compare the two methods blinded for the participants and all health care providers involved in the postoperative care from the time the patient exits the operating room (OR). Blinded studies in surgery are rare but in gastrointestinal surgery, a blinded study of open versus laparoscopic colonic resection has demonstrated to be feasible and thus we believe that such study must be feasible in an RC setting.

Participants will be randomized 1:1 to either ORC or RARC. Blinding: The study is blinded for the patient and for the group of nurses and doctors that will be responsible for the postoperative care. The postoperative care will be managed by members of the bladder cancer team other than the operating surgeon, and OR staff will not be involved in the postoperative care. The abdominal wound will be bandaged to hide the wounds from both an open and laparoscopic procedure. The blinding will be maintained until discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* age> 18
* non-metastatic disease
* fit for both ORC and RARC
* Patient-selected urinary diversion: ileal conduit

Exclusion Criteria:

* if not able to speak/understand Danish
* not able to cooperate for fully informed consent
* need for extensive concomitant surgery (i.e. nephroureterectomy)
* prior down staging chemotherapy (prior neoadjuvant chemotherapy accepted)
* prior radiation therapy
* prior major extensive abdominal or pelvic surgery
* prior peritonitis
* conditions contraindicating extended Trendelenburg's position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Participants blinded at discharge | 12 months
  Number of patients that was not unblinded at discharge

SECONDARY OUTCOMES:
Length of Stay (LOS) | 12 months
  Duration (days) of primary hospitalization. From the date of admission until the date of discharge from hospital.
Days Alive and Out of Hospital (DAOH) | 90 days from surgery
  Number of days alive and out of hospital within 90 days from surgery
30-day complication rate | 30 days after surgery
  Complication rate (Clavien-Dindo)
90-day complication rate | 90 days after surgery
  Complication rate (Clavien-Dindo)
Readmission rate | 90 days after surgery
  Number of readmissions
Quality of Life (QoL): EORTC QLQ-C30 | 90 days after surgery
  Registration of differences in QoL. European Organization for Research and Treatment of Cancer 30-item core quality of life questionnaire (EORTC QLQ-C30 (scale range 0-100, a higher score indicating better quality of life))
Quality of Life (QoL): EORTC QLQ-BLM30 | 90 days after surgery
  Registration of differences in QoL. European Organization for Research and Treatment of Cancer quality of life questionnaire for patients with muscle invasive bladder cancer (QLQ-BLM30 (scale range 0-100, a higher score indicating increase in symptom burden)) will be used.
Blood loss | 4 days after surgery
  Both estimated as well as calculated/hidden blood loss
Use of opioids | until diacharge or up to 90 days, whichever comes first
  Use of opioids, mg total postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maibom SL, Joensen UN, Aasvang EK, Rohrsted M, Thind PO, Bagi P, Kistorp T, Poulsen AM, Salling LN, Kehlet H, Brasso K, Roder MA. Robot-assisted laparoscopic radical cystectomy with intracorporeal ileal conduit diversion versus open radical cystectomy with ileal conduit for bladder cancer in an ERAS setup (BORARC): protocol for a single-centre, double-blinded, randomised feasibility study. Pilot Feasibility Stud. 2023 Jan 13;9(1):7. doi: 10.1186/s40814-022-01229-3. PMID 36639814